CLINICAL TRIAL: NCT06291688
Title: The Efficacy of Applying Mobile Healthcare Education to Improve Cutaneous Self-care Capability for Patients Receiving Targeted Therapy
Brief Title: Applying Mobile Healthcare Education to Improve Cutaneous Self-care Capability
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 202312004RIND
Record Dates: First submitted 2024-02-05; First posted 2024-03-04 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: EGFR Gene Mutation; Drug-Related Side Effects and Adverse Reactions; Cancer, Treatment-Related; Cancer
Keywords: Mobile Healthcare education; Game-based learning; Self-care capability; Learning motivation; Quality of life
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions; Neoplasms, Second Primary; Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Game group (Experimental): An educational game regarding common EGFR-related cutaneous adverse drug reactions on a mobile APP
  Interventions: Behavioral: Mobile healthcare education game
- Text group (Placebo Comparator): An educational text regarding common EGFR-related cutaneous adverse drug reactions on a mobile APP
  Interventions: Behavioral: Mobile healthcare education application

INTERVENTIONS:
Behavioral: Mobile healthcare education game — Game group will download an APP on a smart phone and play the mobile game which contains the educaitonal content regarding EGFR-related cutaneous adverse drug reactions.
  Arms: Game group
Behavioral: Mobile healthcare education application — Text group will download an APP on a smart phone and open the APP to see the text regarding EGFR-related cutaneous adverse drug reactions.
  Arms: Text group

SUMMARY:
The goal of this clinical interventional study is to compare the efficacy of mobile healthcare education in two ways (game-based or text-based) to improve cutaneous self-care capability in cancer patients receiving EGFR-based target therapy. The main questions it aims to answer are:

Impact of different mobile healthcare education ways on cutaneous self-care capability of patients Impact of different mobile healthcare education ways on learning motivation of patients towards cutaneous self-care knowledge and skills

Participants will be randomly divided into two groups. Both groups will download a healthcare education application on their phone. One group will accept the education about the knowledge and self-care skills of cutaneous adverse drug reaction by playing game. In contrast, the other group will accept the same education content by reading text on the phone. Subjects will be asked to use the application at home for two weeks after giving consent to participate this study, and then completed questionnaire three times during study period. The timepoints of completing questionnaire are listed following:

Baseline / pre-intervention test (after signing informed consent form, D1) First post-intervention test (after finishing intervention, D15) Second post-intervention test (D30) Researchers will compare game group and text group to see if game group has better performance on cutaneous self-care capability and learning motivation.

DETAILED DESCRIPTION:
This study is a randomized controlled study. Researchers use a random assignment, parallel two-group pre-test and post-test design to conduct a 1-month interventional study regarding giving health education to patients receiving EGFR-targeted drugs. A total of 3 questionnaires were collected to compare the learning efficacy of giving health education through mobile game and through text. Learning motivation, compliance with prevention care measures, the quality of life and the user experience will be also discussed.

Once the subjects sign the Informed Consent Form, they will be asked to conduct the pre-test questionnaire (D1). Then, the block-randomized assignment will be used to divide subjects into the experimental group or the control group. Both the experimental group and the control group downloaded a health educational APP, regarding cutaneous adverse drug reactions related to EGFR-targeted drugs, on their mobile phones.

After randomization, the researchers will give subjects a randomly generated 4-digit code. Subjects can use this code to log in the APP. After log-in, the subjects in the experimental group will see the interface of an educational game. Meanwhile, the subjects in the control group will see the interface of the text of educational content. Subjects will be asked to play the game or read the text at home for 2 weeks. The subjects will not know the difference between the experimental group and the control group, nor will they know whether they are assigned to the experimental group or the control group, thus maintaining the blindness of the subjects.

After 2 weeks, subjects will be asked to do the first post-test questionnaire (D15) to explore the short-term effect of the APP. Then, they will be encouraged to keep using the APP during the following 2 weeks. At D30, subjects will be asked to do the first post-test questionnaire (D15) to investigate the long-term effect of the APP.

ELIGIBILITY:
Inclusion Criteria:

* Adults whose age is above 18.
* Patients are receiving EGFR-base target drugs now.
* Patients can use smart phone.

Exclusion Criteria:

* Patients with visually impaired, hearing impared or other health related factors cause inability to use smart phone.
* Patients cannot understand study aims and procedures by communicating in Mandarin or Taiwanese.
* Patients cannot follow study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2024-01-26 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the score of cutaneous adverse drug reaction (CADR) knowledge on researcher-designed questionnaire at Day 15 and Day 30. | Day 1, Day 15, Day 30
  Comparing the improvement of CADR knowledge between different groups

SECONDARY OUTCOMES:
Investigate the learning motivation towards CADR by self-designed questionnaire at Day 15 | Day 15
  Compare learning motivations between different groups towards CADR
Change from baseline in the score of the quality of life on DLQI questionnaire at Day 15 and Day 30 | Day 1, Day15, Day 30
  Compare the quality of life between different groups
Investigate the user-experience of the mobile healthcare education APP by researcher-designed questionnaire at Day 15. | Day 15
  Confirm the usability and game-experience of mobile healthcare education APP.
Change from baseline in the score of the self-care measurement adherence on researcher-designed questionnaire at Day 15 and Day30. | Day1, Day15, Day30
  Compare the self-care measurement adherence between different groups

OTHER OUTCOMES:
The correlation among APP usability, learning motivation and self-care capability. | Day 1, Day 15, Day 30
  Investigate the correlation among game usability, learning motivation and self-care capability.

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Chen Chang, Phd, Principal Investigator — National Taiwan University
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No